CLINICAL TRIAL: NCT02807935
Title: The in Vivo Effect of Medical and Surgical Glaucoma Treatments on the Schlemm's Canal
Brief Title: The in Vivo Effect of Medical and Surgical Glaucoma Treatments on the Schlemm's Canal Micro-structure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SHEBA-16-2797-OZ-CTIL
Record Dates: First submitted 2016-06-17; First posted 2016-06-21 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Glaucoma; Cataract
MeSH Terms: conditions — Glaucoma; Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OCT imaging of surgical/pharmacological/laser branch (Other): to evaluate the effect on the conventional outflow pathway, and specifically on the Schlemm's canal (SC) anatomy in the surgical branch:
  1. Before and after trabeculotomy
  2. Before and after cataract surgery
  3. Before and after vitrectomy surgery
  4. Before and after XEN™ Gel Stent implant
  pharmacological branch-
  1. Before and during the treatment with prostaglandins analogs
  2. Before and during the treatment with alpha blockers
  3. Before and during the treatment with beta blockers
  4. Before and during the treatment with carbonic anhydrase inhibitor
  laser branch-
  1. Before and after trabeculoplasty
  2. Before and after laser iridotomy
  3. Before and after yag capsulotomy laser
  Interventions: Device: Optical coherence tomography imaging

INTERVENTIONS:
Device: Optical coherence tomography imaging

SUMMARY:
The purpose of our current series of studies is to evaluate different glaucoma treatments in vivo effect on the conventional outflow pathway, and specifically on the Schlemm's canal (SC) anatomy using Enhanced Depth Imaging (EDI)-optical coherence tomography (OCT) . The images will be taken as part of the patients routine medical follow up (before starting the treatment, and 1,4 and 12 weeks afterwards) diameter, cross-sectional area and volume will be measured using commercially available 3-dimensional reconstruction.

The series of studies will be divided into 3 branches, each branch contains different treatments.For each treatment different patients will be recruited.

The branches are as following-

1. The surgical branch-

   1. Before and after trabeculotomy
   2. Before and after cataract surgery
   3. Before and after vitrectomy surgery
   4. Before and after XEN™ Gel Stent implant
2. The pharmacological branch-

   1. Before and during the treatment with prostaglandins analogs
   2. Before and during the treatment with alpha blockers
   3. Before and during the treatment with beta blockers
   4. Before and during the treatment with carbonic anhydrase inhibitor
3. The laser branch-

   1. Before and after trabeculoplasty
   2. Before and after laser iridotomy
   3. Before and after yag capsulotomy laser

ELIGIBILITY:
Inclusion Criteria:

1. Male or female of any race, at least 18 years of age.
2. Has provided verbal and written informed consent.
3. Able and willing to follow instructions, including participation in all study assessments and visits.
4. Has been referred to one of the treatments mentioned

Exclusion Criteria:

1. Has history of ocular conditions that may affect the SC structure (e.g., ocular neovascularization, anterior segment congenital anomalies)
2. Subject uncooperativeness that restricts adequate examination of IOP, ocular fundus or
3. any ocular or systemic conditions that may reduce OCT image quality (e.g., severe dry eye syndrome, visually significant cataract, limbal opacities, nystagmus, Parkinsonism, etc),
4. Pregnant women or male or female younger than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Mean SC (schlemm's canal) cross-sectional area and volume | 1 year

SECONDARY OUTCOMES:
Correlation of changes with intraocular pressure (IOP) reduction | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- SHEBA medical center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Undecided